CLINICAL TRIAL: NCT02137421
Title: Effects of Resveratrol on Crosstalk Between Canonical β-catenin/Wnt and FOXO Pathways in Coronary Artery Disease Patients With Metabolic Syndrome: A Case Control Study
Brief Title: A Case Control Study of Resveratrol Effects in Coronary Artery Disease Patients With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17001-30-01-91
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2014-05

CONDITIONS: Metabolic Syndrome; Coronary Artery Disease
Keywords: Coronary artery disease; Metabolic syndrome; Resveratrol; β-catenin; Wnt signaling; FOXO; MnSOD
MeSH Terms: conditions — Metabolic Syndrome; Coronary Artery Disease | interventions — Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAD, Metabolic syndrome . (Experimental): Arm1:coronary artery disease with metabolic syndrome . Intervention:Resveratrol (3, 4´, 5 trihydroxystilbene), 50 micromolar,12hour treatment .
  Each experiment repeats three times .
  Interventions: Dietary Supplement: Resveratrol (3, 4´, 5 trihydroxystilbene)
- Healthy subjects . (Experimental): Arm2:healthy subjects Intervention:Resveratrol (3, 4´, 5 trihydroxystilbene), 50 micromolar,12hour treatment .
  Each experiment repeats three times .
  Interventions: Dietary Supplement: Resveratrol (3, 4´, 5 trihydroxystilbene)

INTERVENTIONS:
Dietary Supplement: Resveratrol (3, 4´, 5 trihydroxystilbene) — Resveratrol (RES) (3, 4´, 5 trihydroxystilbene)

SUMMARY:
The aim of this study is to explore the role of Canonical β-catenin/Wnt and forkhead box O (FOXO) pathways by means of investigating their target genes in coronary artery disease (CAD) pathogenesis and to examine the effects of resveratrol (RES) on these pathways in CAD patients.

DETAILED DESCRIPTION:
Metabolic syndrome is a constellation of cardiovascular and metabolic risk factors including obesity, insulin resistance, hypertension and dyslipidemia. Coronary artery disease (CAD) is considerably linked with these risk factors. Oxidative stress has a major role in development of atherosclerosis that is believed as the most common pathologic process underlying CAD. The up-regulated gene-expression of free radical scavenging enzymes such as manganese superoxide dismutase (MnSOD) by members of the forkhead box O (FOXO) transcription factors is considered to be one of the paramount cell defensive mechanisms against oxidative damage. It is now well recognized that β-catenin binds to FOXOs during oxidative stress and acts as the pivotal mediator in canonical Wnt signaling, so that it translocates to the nucleus and interacts with the family of transcription factors T-cell factor/lymphoid enhancer factor (TCF/LEF), to regulate the expression of Wnt target genes. Recent evidence suggested that the canonical Wnt signaling plays a profound role in regulation of lipid metabolism and glucose homeostasis. Peroxisome proliferator-activated receptor delta (PPAR-δ) is one of the Wnt target genes which is believed to be operative in cardiometabolic protection. Interestingly, it has been demonstrated that impaired Wnt signaling pathway is contributed to inflammation, foam cell formation, and endothelial dysfunction which are recognized as atherosclerosis pathogenic factors. Resveratrol (RES) (3, 4´, 5 trihydroxystilbene), a natural polyphenol with antioxidant effects can be found in red grapes and its processed drinks (e.g. red wine), peanuts, pomegranates and mulberries.Increasing body of evidence suggest a protective role for RES against CAD, however the underlying mechanisms still remain to be elucidated. We perform this study on 10 metabolic syndrome patients with three-vessel CAD and 10 sex-aged matched (men with 40-55 years old) healthy subjects as controls. The effects of RES on β-Catenin, manganese superoxide dismutase (MnSOD), and peroxisome proliferator-activated receptor delta (PPAR-δ) expression are evaluated in peripheral blood mononuclear cells (PBMCs) of participants.

ELIGIBILITY:
Inclusion Criteria:

-Three vessel coronary artery disease with metabolic syndrome based on WHO criteria

Exclusion Criteria:

* Malignancy,
* Myocardial infarction,
* Unstable angina,
* Previous coronary intervention,
* Inflammatory diseases,
* Diabetes,
* Hypertension,
* Endocrine disorders,
* Other known chronic diseases,
* Antioxidant therapy or vitamin supplements in the previous 12 months,
* Smokers .

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Relative gene expression by real-time PCR (polymerase chain reaction) | Change from baseline after 12-hour treatment with resveratrol
  PBMCs (2×106/well) are seeded in 96-well plates and undergo overnight incubation in humidified atmosphere at 37° C temperature with 5% CO2(carbon dioxide), then the medium is removed by centrifugation at 300g for 15 min and replaced with a fresh medium containing 50 micromolar resveratrol (dissolved in DMSO (Dimethyl sulfoxide)) for 12 hours. Then, RNA extraction, cDNA(complementary DNA) synthesis and real-time PCR are performed for β-catenin, MnSOD, and PPAR-delta genes .

SECONDARY OUTCOMES:
MnSOD enzyme activity assay . | Change from baseline after 12-hour treatment with resveratrol
Total β-catenin protein measurement | Change from baseline after 12-hour treatment with resveratrol

OTHER OUTCOMES:
PBMCs viability assay by MTT ( 3-(4,5-dimethylthiazol-2-yl)-2,5-diphenyltetrazolium bromide ) test . | Change from baseline after 12 and 24-hour treatment with resveratrol

CONTACTS AND LOCATIONS:
Overall Officials: Taghi Golmohammadi, PhD, Study Chair — Tehran University of Medical Sciences; Arash Hosseinnejad, MD-PhD, Study Chair — Tehran University of Medical Sciences; Reza Meshkani, PhD, Study Director — Tehran University of Medical Sciences; Mahmoud Shirzad, MD, Study Director — Tehran Heart Center,Tehran University of Medical Sciences; Mehrnoosh Shanaki Bavarsad, PhD student, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Islamic Republic of Iran, Tehran, Iran